CLINICAL TRIAL: NCT07030439
Title: An Open-label, Randomized, Single-dose, Two-way Crossover Study to Compare the Bioequivalence of Senaparib 10 mg Capsules Manufactured at Different Manufacturing Sites After Administration in Fasting State in Healthy Chinese Subjects
Brief Title: A Bioequivalence Study to Compare Senaparib Manufactured at 2 Sites in Healthy Subjects in Fasting State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IMP4297-108
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor
MeSH Terms: interventions — senaparib; Long-Term Synaptic Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Senaparib capsules first new manufacturing site then original manufacturing site (Experimental): A single oral dose of 100mg of Senaparib 10 mg strength capsules manufactured by WuXi STA (Wuxi) Co., Ltd. (test product, manufactured at the new manufacturing site) administered in fasting state in first intervention period and then Senaparib 10 mg strength capsules manufactured by WuXi STA (Shanghai) Co., Ltd. (reference product, manufactured at the original manufacturing site) in second intervention period (after washout period: at least 7 days)
  Interventions: Drug: Senaparib 10 mg strength capsules manufactured by WuXi STA (Wuxi) Co., Ltd.; Drug: Senaparib 10 mg strength capsules manufactured by WuXi STA (Shanghai) Co., Ltd.
- Senaparib capsules first original manufacturing site then new manufacturing site (Experimental): A single oral dose of 100mg of Senaparib 10 mg strength capsules manufactured by WuXi STA (Shanghai) Co., Ltd. (reference product, manufactured at the original manufacturing site) administered in fasting state in first intervention period and then Senaparib 10 mg strength capsules manufactured by WuXi STA (Wuxi) Co., Ltd. (test product, manufactured at the new manufacturing site) in second intervention period (after washout period: at least 7 days)
  Interventions: Drug: Senaparib 10 mg strength capsules manufactured by WuXi STA (Wuxi) Co., Ltd.; Drug: Senaparib 10 mg strength capsules manufactured by WuXi STA (Shanghai) Co., Ltd.

INTERVENTIONS:
Drug: Senaparib 10 mg strength capsules manufactured by WuXi STA (Wuxi) Co., Ltd. — A single oral dose of 100mg of Senaparib 10 mg strength capsules manufactured by WuXi STA (Wuxi) Co., Ltd. (test product, manufactured at the new manufacturing site) administered in fasting state in first intervention period and then Senaparib 10 mg strength capsules manufactured by WuXi STA (Shanghai) Co., Ltd. (reference product, manufactured at the original manufacturing site) in second intervention period (after washout period: at least 7 days)
Drug: Senaparib 10 mg strength capsules manufactured by WuXi STA (Shanghai) Co., Ltd. — A single oral dose of 100mg of Senaparib 10 mg strength capsules manufactured by WuXi STA (Shanghai) Co., Ltd. (reference product, manufactured at the original manufacturing site) administered in fasting state in first intervention period and then Senaparib 10 mg strength capsules manufactured by WuXi STA (Wuxi) Co., Ltd. (test product, manufactured at the new manufacturing site) in second intervention period (after washout period: at least 7 days)

SUMMARY:
An Open-label, Randomized, Single-dose, Two-way Crossover Study to Compare the Bioequivalence of Senaparib 10 mg Capsules Manufactured at Different Manufacturing Sites After Administration in Fasting State in Healthy Chinese Subjects

DETAILED DESCRIPTION:
An Open-label, Randomized, Single-dose, Two-way Crossover Study to Compare the Bioequivalence of Senaparib 10 mg Capsules Manufactured at Different Manufacturing Sites After Administration in Fasting State in Healthy Chinese Subjects.

32 Subjects are planned to be enrolled. At least, 26 subjects are planned to be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understood the purpose, nature, methods and possible adverse reactions of the trial, voluntarily participated in the trial, and signed an informed consent form before any trial procedure, and promised to participate in all procedure of the trial.
2. Healthy Chinese male subjects aged 18 to 55 (inclusive) at screening.
3. Body mass index (BMI) ranged from 19.0 to 26.0 kg/m2 (inclusive); body weight ≥ 50.0 kg.
4. Subjects could communicate well with the investigators and understood and abided by the requirements of this trial.

Exclusion Criteria:

1. Subjects with diseases with clinical abnormality, including but not limited to disease concerning nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolic system and skeletal system.
2. Subjects with allergic history (including drug and food allergies, etc.).
3. Subjects with history of dysphagia or any gastrointestinal disease that affected drug absorption judged by the investigator.
4. Subjects who had received surgery within 3 months before screening, or planned to have surgery during the trial, or those who had previous surgery that would affect drug absorption (e.g. gastrectomy).
5. Subjects who could not tolerate venipuncture, or had a history of needlesickness and fainting at the sight of blood.
6. Subject with lactose intolerability (who having had milk diarrhea).
7. Subjects who had drug abuse history within 6 months before screening, or had a positive urine drug screening (screening or baseline period) result.
8. Subjects who consumed more than 14 units of alcohol per week (1 unit of alcohol = 360 mL beer, 150 mL wine, or 45 mL liquor) within 3 months before screening, or who had a positive result of alcohol breath test (screening or baseline period), or could not give up alcohol during the trial.
9. Subjects who consumed an average of more than 5 cigarettes per day within 3 months before screening, or who could not stop using any tobacco products during the trial.
10. Subjects who consumed an average of excessive amounts of tea, coffee and / or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) every day within 3 months before screening.
11. Subjects who had participated in clinical trials of other study drugs/devices within 3 months before the first dose of the investigational drug, or had participated in 3 or more clinical trials of drugs/devices in the past year; if other study drugs had a longer half-life, the time interval would be longer and was required to be 5 half-lives of the drug.
12. Subjects who donated blood including blood component or had massive blood loss (≥ 200 mL), or received blood transfusion or used blood products and blood biological products within 3 months before screening.
13. Subjects who received live vaccines within 4 weeks before screening.
14. Subjects who had taken any drugs [such as: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; SSRI(selective serotonin reuptake inhibitor) antidepressants, cimetidine, macrolides, sedative hypnotics, antihistamines, antivirals (such as saquinavir), calcium antagonists (such as diltiazem, verapamil), rifamycins (such as rifampicin)] that potently inhibit or induce CYP3A4 enzymes within 28 days before the use of the investigational drug. If the past drug used had a longer half-life, the time interval would be longer and was required to be 5 half-lives of the drug, e.g., phenobarbital required a 5-week washout period.
15. Subjects who had taken prescription drugs, over-the-counter drugs, dietary supplements or Chinese herbal medicine within 14 days before the first dose of the investigational drug. If the past drug used had a longer half-life, the time interval would be longer and was required to be 5 half-lives of the drug. Limited use of over-the-counter drugs that were not considered to affect the overall outcome of the study was allowed on a case-bycase basis after approval by the sponsor and the investigator.
16. Any test result of hepatitis B surface antigen, hepatitis B core antibody, hepatitis C virus antibody, human immunodeficiency virus (HIV) antibody, or treponema pallidum antibody was positive.
17. At screening, vital signs (blood pressure, pulse and body temperature) examination, comprehensive physical examination and laboratory tests (hematology, blood biochemistry, urinalysis) indicated abnormal results with clinical significance according to the investigator. The reference normal range of vital signs (including the cut-off value) was as follows: Sitting systolic blood pressure was 90 to 140 mmHg, diastolic blood pressure was 60 to 90 mmHg, pulse was 60 to 100 bpm, body temperature (ear temperature) was 35.7 to 37.9°C. The specific situation was comprehensively determined by the investigator.
18. At screening, the corrected QT interval (corrected by Fridericia's formula, QTcF = QT/RR1/3) > 450 msec or QRS complex > 120 msec was obtained by 12-lead ECG in supine position in resting state (at least 5 min). If QTc was more than 450 msec or QRS was more than 120 msec, ECG measurement should be repeated twice, and the average value of QTc or QRS measured three times was judged by the investigator as abnormality with clinical significance.
19. Subjects who were allergic to Senaparib, or to any ingredients of the preparation.
20. Vigorous exercise could not be avoided within 48 h before the first dose of the investigational drug and during the trial.
21. Subjects who consumed any food or beverages containing alcohol, caffeine, chocolate, or rich in xanthine within 48 h before the first dose of the investigational drug; or those who could not abstain from these products during the trial.
22. Subjects who could not abstain from grapefruit or grapefruit-related citrus (eg, pomelo) or juice within 7 days before the first dose of investigational drug and during the trial.
23. Subjects or its partners who had birth plan, or were unwilling to adopt effective contraception methods, or had sperm donation plan throughout the trial and within 90 days after the last dose of the investigational drug.
24. Subjects who were unwilling or unable to follow the lifestyle guidelines described in the study protocol (such as dietary restrictions and activity requirements).
25. Subjects who had other acute or chronic medical or psychiatric diseases, which may increase the risks of participating in this trial, or may interfere with the interpretation of the trial results, were judged unsuitable to participate in this trial by the investigator.
26. Subjects judged by the investigator to be unsuitable for participation in the trial.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-07-18 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-72 hour
  Maximum concentration
AUC0-last | 0-72 hour
  Area under the curve from time 0 to the last time with quantifiable concentration
AUC0-inf | 0-72 hour
  If the data were available, area under the curve from time 0 to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Chuanling Li, Principal Investigator — Xuzhou Central Hospital
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No